CLINICAL TRIAL: NCT00507000
Title: Role of Oral Vitamin D as an Adjunct Therapy in Category I Pulmonary Tuberculosis Along With Assessment of Immunological Parameters. (Double-blind, Randomized, Placebo-Controlled, Clinical Trial)
Brief Title: Pulmonary Tuberculosis and Vitamin D
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indian Council of Medical Research (Other Government)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Depratment of Biotechnology (Dr R Goswami, Principal Investigator), All India Institute of Medical sciences, New delhi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BT/pr7898/Med/14/1179/2006
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2009-07

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A, Cholecalciferol (Active Comparator): A Cholecalciferol Drug: Cholecalciferol 60,000 IU sachet and calcium carbonate Oral cholecalciferol (vitamin D)60,000 IU weekly along with daily oral dose of 1 gm calcium carbonate for first two months followed by 1 gm of elemental calcium in form of calcium carbonate daily cholecalciferol (vitamin D)60,000 IU per month for the next four months
  Interventions: Drug: Cholecalciferol
- Vitamin D and Tuberculosis (Placebo Comparator): B, Lactose
  Interventions: Drug: Lactose granules

INTERVENTIONS:
Drug: Cholecalciferol — Drug: Cholecalciferol Drug: Cholecalciferol 60,000 IU sachet and calcium carbonate Oral cholecalciferol (vitamin D)60,000 IU weekly along with daily oral dose of 1 gm calcium carbonate for first two months followed by 1 gm of elemental calcium in form of calcium carbonate daily cholecalciferol (vitamin D)60,000 IU per month for the next four months Arms: A, Cholecalciferol
  Other Names: Vitamin D
  Arms: A, Cholecalciferol
Drug: Lactose granules — Drug: Lactose placebo Lactose placebo granules in identical sachet given weekly and two lactose tablets for first two months followed one sachet of placebo granules every month and two tablets of lactose containing placebo tablets taken daily for next four months
  Arms: Vitamin D and Tuberculosis

SUMMARY:
Tuberculosis and vitamin D deficiency are important public health problems in India. Before the advent of effective antitubercular therapy, patients with tuberculosis were advised treatment and rest at sanatorium where sunshine was available in plenty. There have been reports associating vitamin D deficiency with tuberculosis in terms of incidence and beneficial response following addition of vitamin D to antitubercular therapy. Sputum AFB conversion rate is higher in patients with tuberculosis supplemented with vitamin D. The present study would systematically assess role of adjunct vitamin D therapy (cholecalciferol) in patients with pulmonary tuberculosis.

DETAILED DESCRIPTION:
Tuberculosis and vitamin D deficiency are important public health problems in India. In recently published studies from our center, up to 90% of the apparently healthy subjects in Delhi were classified either as as vitamin D insufficient or deficient by using serum 25(OH)D cut off levels of 20 ng/ml and 32 ng/ml respectively. Before the advent of effective antitubercular therapy, patients with tuberculosis were advised treatment and rest at sanatorium where sunshine was available in plenty. In the western literature, there have been reports associating vitamin D deficiency with tuberculosis in terms of incidence and beneficial response following addition of vitamin D to antitubercular therapy. A few pilot studies have shown that sputum conversion rate is higher in patients with tuberculosis supplemented with vitamin D.

In the above context the mechanisms linking vitamin D deficiency and its effect on tuberculosis are currently under investigation. In order to understand the link two types of studies have been conducted (a) clinical studies associating vitamin D deficiency and tuberculosis and (b) in-vitro assessment of molecular immune changes related to vitamin D exposure. With the currently available knowledge, the linkage between the two disorders is being explained by the broad role of vitamin D deficiency in modulation of cell-mediated immunity.

Patients with military tuberculosis are characterized by decreased levels of Th1 cytokines and increased levels of IL-10 compared with the healthy infected and noninfected controls. Current literature suggests that long-term control of M. tuberculosis infection is associated with elevated Th1 responses and concomitant inhibition of the Th2 response

Peripheral blood mononuclear cells have been shown to express vitamin D receptors. Incubation of macro¬phages with physio¬logical concentration of 1,25 (OH)D [10-9M] results in inhibition of intracellular growth of Mycobacterium tuberculosis. 1,25-dihydroxycholecalciferol, has significant immunomodulatory effects leading to (a) shift in cytokine profile of T-helper (Th1 to Th2) and (b) reduced antigen presentation, reduced production of Th1-promoting cytokines, reduced expression of co-stimulatory molecules in the antigen-presenting cell. In addition, it was demonstrated that the addition of vitamin D3 derivatives inhibits the differentiation of IFN-gamma-producing Th1 cells while it augments the differentiation of IL-4- or IL-10-producing Th2 cells.

There are no systematic data from our country assessing association between vitamin D deficiency and tuberculosis and the possible role of vitamin D related modulation in the tuberculosis specific cellular immune response. The present study has been planned with the following hypothesis

Hypothesis: Patients with pulmonary tuberculosis and vitamin D deficiency when treated with vitamin and antitubercular therapy are likely to show early sputum conversion and immune response favoring resolution of tuberculosis

ELIGIBILITY:
Inclusion Criteria:

1. All patients of either sex with Newly diagnosed sputum positive pulmonary TB cases
2. Aged between 18 to 60 yrs

Exclusion Criteria:

1. Category II pulmonary TB and multi-drug resistant TB (MDR-TB) patients
2. Presence of secondary immunodeficiency states : HIV, organ transplantation, diabetes mellitus, malignancy, treatment with corticosteroids
3. Hepatitis B and C positivity
4. Patients with extrapulmonary TB and/or patients requiring surgical intervention
5. Currently receiving cytotoxic therapy, or have received it within the last 3 months
6. Pregnancy and lactation
7. Patients with a known seizure disorder
8. Patients with known symptomatic cardiac disease, such as arrhythmias or coronary artery disease
9. Patients with abnormal renal functions (serum creatinine more than 2 mg/dl; more than 2+ proteinuria)
10. Patients with abnormal hepatic functions (bilirubin = 1.5 mg/dl; AST, ALT, SAP > 1.5 times above upper limit
11. Patients with hematological abnormalities (WBC lesser than or equal to 3000/mm3; platelet count less than or equal to 100,000/mm3)
12. Seriously ill and moribund patients with complications : tachypnoea, chronic cor pulmonale, congestive cardiac failure, BMI<15, severe hypoalbuminemia
13. Patients unable to comply with the treatment regimen
14. Patients with history of alcohol or drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Time to convert from sputum positivity to negativity | Two months after the last recruitment

SECONDARY OUTCOMES:
1 To study the relapse rate and safety assessment 2 To study the effect of Vitamin D supplementation on the pattern of effector immune function in patients suffering from pulmonary Tuberculosis. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Goswami, MD, DM, Principal Investigator — Associate Professor, Depratment of Endocrinology and Metabolism, All India Institute of Medical Sciences, New delhi 110029; SK Sharma, MD, PHD, Principal Investigator — Head, Depratment of Medicine, All India Institute of Medical Sciences, New Delhi 110029; DK Mitra, MBBS, PhD, Principal Investigator — Associate professor, Department of Transplant immunology and immunogenetics, All India Institute of Medicasl Sciences, New delhi 110029, India; Urvashi B Singh, MD, PhD, Principal Investigator — Assistant Professor, Deprtament of Microbiology, All India Institute of Medical Sciences, new delhi 110029; Nandita Gupta, PhD, Principal Investigator — Additional Porfessor, Department of Endocrinology and Metabolism, All India Institute of Medical Sciences, New Delhi 110029, India; Bindu Dey, PhD., Study Director — Adviser, Department of Biotechnology, Lodhi Road, New Delhi-110003, India
Locations (1):
- Depratment of Endocrinology;Medicine, All India Institute of Medical sciences, and DBT, Delhi, New Delhi, India